CLINICAL TRIAL: NCT04629092
Title: The Effect of Upper Limbs Motion on Lower Limb Biomechanics and Muscle Activity During Single-leg Jump Landing After Anterior Cruciate Ligament Reconstruction
Brief Title: The Effect of Upper Limbs Motion During Single-leg Jump Landing After Anterior Cruciate Ligament Reconstruction
Status: Completed | Type: Observational
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Other Study IDs: YM108023E
Record Dates: First submitted 2019-08-15; First posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2019-05

CONDITIONS: Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate the effect of upper limbs motion on lower limb biomechanics and muscle activity during single-leg jump landing after anterior cruciate ligament reconstruction.

DETAILED DESCRIPTION:
More and more people join in different sports in recent years. But the incidence of sports injury also increases. And the most frequently occurring and debilitating knee injury in sports is rupture of the anterior cruciate ligament (ACL). Patients who aim to return to their preinjury sports should undergo anterior cruciate ligament reconstruction (ACLR) in order to maximize knee stability. The overall incidence rate of a second ACL injury within 24 months after ACLR was nearly 6 times greater than that in healthy participants. Although many studies have showed about biomechanical and neuromuscular risk factors during jump landing which were thought to associate with the secondary injury after ACLR, these studies all focused on the motion of lower extremity. But actually, people often use their upper limbs to catch or throw a ball during jump landing in playground. Whether the upper limbs motion will affect the muscle coordination of lower extremity during jump landing is still unknown. Therefore, the purpose of our study is to investigate the effect of upper limbs motion during single-leg jump landing after ACLR.

ELIGIBILITY:
Inclusion Criteria:

* Only one leg has operation of ACL reconstruction
* At least 1 year after ACLR or have been back to sports
* Exercise in sports regularly.

Exclusion Criteria:

* Other operation of lower extremity exclude ACLR
* Any diseases or poor condition that will affect jumping or deterioration after jumping.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Age between 20-50 years old
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Kinematics of lower-limb during landing phase | from taking off to landing, about 5 seconds.
  The data will be collected by VICON motion capture system, include hip, knee and ankle joint angle in three plane. (frontal plane, sagittal plane and transverse plane)
Kinetics of knee joint during landing phase | from taking off to landing, about 5 seconds.
  The data will be collected by VICON motion capture system and calculated by inverse dynamics, include knee flexion/extension moment, abduction/adduction moment, internal/external rotation moment.
Muscle onset time of lower-limb muscles during landing phase | from taking off to landing, about 5 seconds.
  The data will be collected by wireless electromyography, include rectus femoris, vastus medialis, vastus lateralis, biceps femoris, semitendinosus.
Muscle activation of lower-limb muscles during landing phase | from taking off to landing, about 5 seconds.
  The data will be collected by wireless electromyography, include rectus femoris, vastus medialis, vastus lateralis, biceps femoris, semitendinosus, anterior tibialis, medial gastrocnemius
Muscle activation-Hamstring and Quadriceps ratio (H/Q ratio) during landing phase | from taking off to landing, about 5 seconds.
  The data will use the amount of hamstring and quadriceps muscle activation to calculate H/Q ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Wei Chou, PhD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang-Ming University, Taipei, Taiwan